CLINICAL TRIAL: NCT07377396
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Ascending Doses of ARGX-124 in Healthy Adult Participants
Brief Title: A Study to Assess the Safety of ARGX-124 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-124-1-HV-1001
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARGX-124 (Experimental): Participants receiving the experimental drug
  Interventions: Biological: ARGX-124
- Placebo (Placebo Comparator): Participants receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARGX-124 — Administrations of ARGX-124
  Arms: ARGX-124
Other: Placebo — Administrations of placebo comparator
  Arms: Placebo

SUMMARY:
This study aims to assess the safety of ARGX-124 in healthy adults. Another aim is to measure the amount of ARGX-124 in the blood over time to learn how it acts and moves in the body and how the immune system responds to it. Participants will remain in the study for up to approximately 23 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the local legal age of consent and aged 18 to 65 years, inclusive, when signing the ICF.
* Is a female of Nonchildbearing Potential (postmenopausal or surgically sterilized) or a male.
* Has a body weight between 50 and 120 kg and a BMI between 18 and 30.5 kg/m2, inclusive.

Exclusion Criteria:

* Has any current or past clinically meaningful medical or psychiatric condition that, in the investigator's opinion, would confound the study results or put the participant at undue risk.
* Has IgG levels <6.0 g/L at screening.
* Has a history of an immunosuppressive disease or an immunosuppressive condition at screening.
* Previously participated in an ARGX-124, ARGX-213, or efgartigimod clinical study and received at least 1 dose of the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs and AEs leading to ARGX-124 discontinuation | Up to 23 weeks
  AE : adverse event ; SAE : serious adverse event.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 23 weeks
Percent change from baseline in total IgG levels in serum over time | Up to 23 weeks
  IgG : immunoglobulin G
Incidence of ADA against ARGX-124 in serum | Up to 23 weeks
  ADA : anti-drug antibodies

IPD SHARING:
Plan to Share IPD: No